CLINICAL TRIAL: NCT03675425
Title: Chest Shielding for Prevention of a Patent Ductus Arteriosus in Preterm Infants Receiving Phototherapy Effect of Phototherapy
Brief Title: The Effects of Phototherapy in Preterm Infants Pda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 148/2017
Record Dates: First submitted 2018-07-15; First posted 2018-09-18 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-07

CONDITIONS: Patent Ductus Arteriosus After Premature Birth; Hyper Bilirubinemia
Keywords: Chest shielding; Patent Ductus Arteriosus; Chest Childing
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: non chest shielding (Experimental): non chest shielding generic name: non dosage: non frequency and duration: in first 48 h eco with pad diameter will be measured in before and after phototherapy,
  Interventions: Other: Group 1: non chest shielding
- Group 2: chest shielding (Placebo Comparator): chest shielding generic name: Phototrephy dosage: non frequency and duration: in first 48 h echo with pad diameter will be measured in before and after phototherapy,
  Interventions: Other: Group 2: chest shielding

INTERVENTIONS:
Other: Group 1: non chest shielding — non chest childin: infants will be randomized into two different phototherapy groups eco with pad diameter will be measured in before and after phototherapy,
  Arms: Group 1: non chest shielding
Other: Group 2: chest shielding — chest childing: infants will be randomized into two different phototherapy groups eco with pad diameter will be measured in before and after phototherapy,
  Arms: Group 2: chest shielding

SUMMARY:
The study was designed to assess whether chest shielding during phototherapy reduces the incidence of PDA, as assessed by serial echocardiographic examinations, in a population of extremely preterm infants born at lower 30 week gestation.

DETAILED DESCRIPTION:
Phototherapy is a therapeutic intervention frequently used for management of neonatal hyperbilirubinaemia in extremely premature infants, especially in the first week when patency of the ductus is a clinical problem. Phototherapy has also been implicated in increased ductal patency. One randomized, controlled trial showed that chest shielding during phototherapy reduced the incidence and severity of PDA by 50% in preterm infants. These findings were mainly based on clinical evaluation of the ductus with echocardiographic studies performed only on a subgroup of infants noted to have a murmur on clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* Gestational week ≤ 30 weeks receiving phototherapy due to jaundice and infants who can perform echocardiography before and after treatment will be included in the study.

Exclusion Criteria:

* Babies with congenital heart disease.
* Infants with major structural anomalies and infants who can not undergo echocardiography before or after treatment.

Ages: 3 Days to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2018-07-08 (Actual); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
echocardiographic examination | first week
  presence of Patent Ductus arteriozus

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Alyamaç Dizdar, MD, Study Director — zekai tahir burak matarnity teaching hospital
Locations (1):
- Zekai Tahir Burak Matarnity Teaching, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided